CLINICAL TRIAL: NCT03035695
Title: Pre Hospital Hemorrhagic Control Effectiveness of Axiostat® Dressing Versus Conventional Method in Acute Hemorrhage Due to Trauma
Brief Title: Studying Safety & Efficacy of Axiostat® Dressing in Acute Hemorrhage Due to Trauma-Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Axio Biosolutions Pvt. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABPL/003
Record Dates: First submitted 2017-01-23; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Bleeding
Keywords: Trauma; Scalp injuries; Profused Bleeding; Accident
MeSH Terms: conditions — Hemorrhage; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Axiostat® Size (Experimental): Device: Axiostat® Size: 8 x 5 cm Axiostat® is a sterile, non-absorbable haemostatic dressing intended to control profuse bleeding within minutes of application by providing an active mechanical barrier to the wound site.
  Mechanism of action is such that Axiostat® is an extremely positive dressing that becomes very sticky in the presence of negatively charged blood and thus seals the wound area.
  Interventions: Device: Axiostat®
- Cotton Gauze (Active Comparator): Cotton Gauze Size: 8 x 5 cm
  Interventions: Device: Cotton Gauze

INTERVENTIONS:
Device: Axiostat®
  Other Names: Haemostatic dressing
  Arms: Axiostat® Size
Device: Cotton Gauze
  Arms: Cotton Gauze

SUMMARY:
The aim of this study was to evaluate the efficacy and safety to use external haemostatic between Axiostat® (Chitosan haemostatic dressing) and conventional cotton gauze dressing as a pre hospital acute hemorrhagic control in trauma in ambulance settings.

DETAILED DESCRIPTION:
Abstract:

Accidents and trauma comprise leading causes of death and disability throughout the world. In developing countries such as India, where emergency trauma care is still in its infancy, it accounts for almost 10% deaths every year. Lack of adequate pre-hospital care and uncontrolled bleeding from wound site are stated to be the prominent reasons for such deaths.

In this study, a novel chitosan-based haemostatic dressing (Axiostat®, Axio Biosolutions, India) was investigated as an initial hemorrhage controlling device in pre-hospital scenario. The study was conducted with the help of 35 Emergency Medical Technicians (EMTs).

A total of 133 patients with scalp wound injury were identified for the study, of which 104 patients meeting the selection criteria were included in the study. The selected patients were randomly assigned into two groups, the test group consisting of 47 subjects received Axiostat® treatment; whereas, 57 subjects in the control group were treated with a conventional cotton-gauze dressing. All subjects needed suturing as the subjects included in the study were brought with open scalp wounds.

The Axiostat® showed a superior efficacy in controlling bleeding in comparison to the cotton gauze. The average time for haemostasis with cotton gauze dressing was about 18.56 ± 5.04 minutes; while with Axiostat® haemostasis was achieved in less than 5 minutes (4.68 ± 1.04 min).

On analyzing this study, it was evident that Axiostat® dressing enables early haemostasis which prevents much blood loss and the wound becomes very clean on removal of dressing for later wound suturing when compared to normal cotton gauze.

These findings demonstrated the potential of Axiostat® as a first-line intervention in controlling acute hemorrhage in the pre-hospital scenarios.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Patient and/or patient's legal representative and/or impartial witness have been informed of the nature of the study and agree to its provisions and have provided written informed consent as approved by the IEC of MIMS, Kerala, India.
* Patients with bleeding wounds over scalp which can due to any injury.
* The wounds must be bleeding at the time of baseline assessment.
* The targeted wound size should be such that it should be covered by single available size of the study device as per the instructions for use.

Exclusion Criteria:

* The exclusion criteria for the study involved prior diagnosis of disease or medical condition affecting the ability of blood to clot (e.g., hemophilia).
* A non-survivable injury as per the investigators' discretion.
* Patients who in the opinion of the investigator may not complete the study for any reason, e.g. Patients requiring immediate suturing. Grossly infected wounds that may reasonably be expected to require multiple debridement procedures prior to clearance of bacteria and non-viable tissue from the wound, in case of old wound.
* Patient is currently participating in an investigational drug or device study that has not yet completed its primary endpoint or interferes with procedure and assessments in this trial.
* Patients with Surgical/iatrogenic wound.
* Patients with a major head injury, spinal injury, neck injury, abdominal injury, deep wound injury, fracture, hemorrhagic shock, foreign materials inside the wound like stab injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Time to achieve hemostasis | 1 Day
  Time to achieve hemostasis by observing the time at which blood oozing through or from periphery of the dressing stops.

SECONDARY OUTCOMES:
Number of patients with rebleeding | 1 Day
  Number of patients with rebleeding will be counted (unit of measurement is number/count of patients)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mohmmad Kabeer, Principal Investigator — Malabar Institute of Medical Sciences
Locations (1):
- Malabar Insitute of Medical Sciences, Calicut, Kerala, India

IPD SHARING:
Plan to Share IPD: No